CLINICAL TRIAL: NCT06225986
Title: The Living Memory Home: Reducing Grief and Improving Relationships Between Home-Based Patients With ADRD and Their Family Caregivers
Brief Title: Living Memory Home-4-Dementia Care Pairs
Acronym: LMH-4-DCP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 23-07026251; R21AG077144 (NIH)
Record Dates: First submitted 2024-01-09; First posted 2024-01-26 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Dyadic Family Caregiver-person With Dementia Online Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LMH-4-DCP Intervention (Experimental)
  Interventions: Behavioral: LMH-4-DCP
- Attention Control Arm (Active Comparator)
  Interventions: Behavioral: LMH-4-DCP access without reminiscence activities

INTERVENTIONS:
Behavioral: LMH-4-DCP — Reminiscence-based intervention for family caregiver-Persons with Dementia (PwD) dyads to record and reflect on meaningful memories to address family caregivers' pre-loss grief and enhance relationship quality.
  Arms: LMH-4-DCP Intervention
Behavioral: LMH-4-DCP access without reminiscence activities — Participants in the attention control condition will have access to a version of LMH-4-DCP excluding reminiscence-specific activities.
  Arms: Attention Control Arm

SUMMARY:
The purpose of this study is to evaluate an online platform -- the Living Memory Home for Dementia Care Pairs (LMH-4-DCP) for persons with dementia and their family caregivers to engage in reminiscence activities together and record meaningful memories.

The main aims of this study are:

* To evaluate the feasibility and acceptability of the LMH-4-DCP platform.
* To explore the potential for LMH-4-DCP to reduce feelings of pre-loss grief and enhancing relationship quality in dementia family caregivers and their care-recipients ('Care-Pairs')

Care pair participants will be asked to log-in to LMH-4-DCP and complete study activities three times per week for two weeks. Researchers will compare the intervention group to an attention control condition to see if LMH-4-DCP's use is associated with reduced feelings of caregiver pre-loss grief and improved care pair relationship quality at follow-up.

DETAILED DESCRIPTION:
The goal of this randomized controlled trial is to evaluate the Living Memory Home for Dementia Care Pairs (LMH-4-DCP) web application, a dyadic online psychosocial reminiscence platform, to reduce feelings of pre-loss grief and improve relationship quality in individuals with dementia and their family caregivers ('Care Pairs').

The main aims of this study are:

* To evaluate the feasibility and acceptability of the LMH-4-DCP platform.
* To explore the influence of the LMH-4-DCP intervention on reducing feelings of pre-loss grief and enhancing relationship quality in the care pair

Caregiver participants randomized to the intervention condition will be asked to log-in to LMH-4-DCP and complete reminiscence activities three times per week for two weeks. Researchers will compare the intervention group to an attention control condition, which includes LMH-4-DCP use without reminiscence-specific features, to see if LMH-4-DCP's use is associated with reduced feelings of caregiver pre-loss grief and improved care pair relationship quality at follow-up.

ELIGIBILITY:
Inclusion Criteria:

Family Caregivers:

* be a primary source of care for a family member in the early to moderate stages of dementia
* 18 years of age or older
* English-speaking
* able to use the internet and has internet access
* residing in the United States

Exclusion Criteria:

Caregiver exclusion criteria:

* is not the primary family caregiver of the PwD
* under the age of 18-years-old
* exhibits cognitive impairment (by scoring 3 or more on the SPMSQ)
* does not speak English as a primary language.

PwD exclusion criteria:

* severe cognitive impairment detected by the clinical or study staff using validated, brief screening tools (e.g., a score of 8 errors or more on the SPMSQ)
* does not demonstrate capacity to consent (e.g., a score of 9 or fewer errors on the University of California-San Diego Brief Assessment of Capacity to consent
* PwD is living in a long-term care facility
* does not speak English as a primary language
* is under the age of 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2025-06-16 (Estimated); Study Completion 2025-06-16 (Estimated)

PRIMARY OUTCOMES:
The Feasibility of the LMH-4-DCP application as measured by the number of website logins per participant out of total required (minimum= 6). | 2 Weeks
  The feasibility of the application will be measured by the number of times the participant logs in to the LMH-4-DCP web application. The minimum number of logins recommended to the participants is 6.
The Feasibility of the LMH-4-DCP study as measured by participant retention, as indicated by the number of participants lost to follow-up. | 2 Weeks
  Participant retention, as an aspect of feasibility, will be measured by the recorded number of participants number lost to follow-up. A number of the enrolled participants who the study team contacted three times, but did not answer or continue participation, will be recorded.
The Feasibility of the LMH-4-DCP study as measured by participant retention, as indicated by the number of recorded dropouts. | 2 Weeks
  Participant retention, as an aspect of feasibility, will be measured by the recorded number of dropouts. A number of the participants who asked to withdraw/drop-out from the study after being enrolled will be recorded.
The Feasibility of the LMH-4-DCP application as measured by the time spent in each activity within the web application. | 2 Weeks
  The feasibility of the application will be measured by the time spent in each activity. The time will be measured in minutes and seconds. For example, 5 minutes and 30 seconds.
The Feasibility of the LMH-4-DCP study as measured by the proportion of family caregivers who (1) consent to participate. | 2 Weeks
  The feasibility of the LMH-4-DCP study will be measured by the proportion of family caregivers who consent to participate among those who were invited and screened into the study.
The Feasibility of the LMH-4-DCP study as measured by recruitment rates and the proportion of family caregivers (2) decline participation. | 2 Weeks
  The feasibility of the LMH-4-DCP study will be measured by the proportion of family caregivers who decline to participate among those who were invited and screened into the study.
The Feasibility of the LMH-4-DCP study as measured by recruitment rates and the proportion of (3) are deemed ineligible based on screening criteria. | 2 Weeks
  The feasibility of the LMH-4-DCP study will be measured by the proportion of family caregivers who are deemed ineligible based on screening criteria among those who were invited to participate in the study.
The Usability of the LMH-4-DCP application as measured by the System Usability Scale (SUS). | 2 Weeks
  The usability of the web application will be measured by the SUS. This scale is a 10-item assessment of the usability of a system, helping identify areas for improvement. Response options range from 1=Strongly Disagree to 5-Strongly Agree. Scores range from 0-100, with higher scores indicative of greater usability.
The Acceptability of the LMH-4-DCP application as measured by a survey that measures the participants satisfaction and acceptability of the application. | 2 Weeks
  The acceptability of the web application will be measured by the use of surveys assessing usability, engagement, acceptability, suggestions for improvement.
  Participants will be asked to rate their agreement with statements including "I enjoyed my experience using the LMH-4-DCP application". Response options are rated on a five-point scale from 1-Strongly Disagree to 5-Strongly Agree.
  Because the surveys differ slightly by group, the intervention groups scores range from 8-40 and the control groups' scores range from 7-35, with higher scores indicating greater satisfaction and acceptability.
The Acceptability of the LMH-4-DCP application as measured by a qualitative survey that measures the participants satisfaction and acceptability of the application. | 2 Weeks
  The acceptability of the web application will be measured by the use of open-ended items assessing usability, engagement, acceptability, suggestions for improvement.
  The intervention group participants will also be administered five open-ended qualitative items asking for feedback on LMH-4-DCP. Sample items include: "Which LMH-4-DCP features were most valuable and why?"

SECONDARY OUTCOMES:
Change in Grief Severity as measured by the Pre-Loss Grief-12 (PG-12) | Baseline, 2 Weeks
  Caregivers' pre-loss grief assessed using the validated 12-item PG-12-R instrument; Scores ranging from 12-60, with higher scores indicative of greater feelings of pre-loss grief.
Change in Relationship Quality as measured by the Relational Deprivation Scale. | Baseline, 2 Weeks
  The first measure of relationship quality will be the validated six-item Relational Deprivation Scale, which measures the perceived loss of relationship as a result of the care-recipient's illness. Response options range from 1=Not at all to 4=Completely. Scores range from 6 to 24, with higher scores indicative of poorer relational quality.
Change in Relationship Quality as measured by the Mutuality Scale. | Baseline, 2 Weeks
  The second measure of relationship quality will be the validated 15-item Mutuality Scale, which measures the extent of positive aspects of caregiving. Response options range from 0=Not at all to 4=A Great Deal. Scores range from 0-60, with higher scores reflecting greater levels of mutuality.
Change in Relationship Quality as measured by the Relationship Rewards Scale (RSS) Scale. | Baseline, 2 Weeks
  The third measure of relationship quality will be the eight-item validated RSS, where the caregiver reports experiences of relationship quality before and after the care-recipient's diagnosis. Responses range from 1=Never to 4=Always. Scores range from 8-32, with higher scores indicating greater relational quality.

CONTACTS AND LOCATIONS:
Overall Officials: Holly Prigerson, PhD, Principal Investigator — Weill Medical College of Cornell University; Francesca Falzarano, PhD, Principal Investigator — University of Southern California; Weill Cornell Medicine
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected for the LMH-4-Dementia Care Pairs study will only be shared after we have published the data addressing the study's specific aims. Intellectual property and data generated under this project will be administered in accordance with both Weill Cornell Medicine (WCM) and NIH policies, including the NIH Data Sharing Policy and Implementation Guidance. After publication of our main findings, access to databases and associated software tools generated and the code to create these tools under the project will be available for educational, research and non-profit purposes.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: These data will be shared after we have published the specific aims of this study. Requests for the code used to create LMH-4-Dementia Care Pairs will be reviewed by the investigative team and shared once we have published the findings showing it is safe and therapeutic.
Access Criteria: 1) to use the data for research purposes only; 2) not to identify any individual participant; 3) to secure the data using appropriate computer technology such as password-protected servers and files; and 4) to return and/or destroy data after analyses are complete.